CLINICAL TRIAL: NCT02765061
Title: Hyponatremia and Hypoalbuminemia is Morbimortality Predictors in Coronary Artery Bypass
Brief Title: Hyponatremia and Hypoalbuminemia is Morbimortality Predictors in Coronary Artery Bypass Graft Surgery
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Ankara University, Ankara University
Other Study IDs: TYİH
Record Dates: First submitted 2016-05-05; First posted 2016-05-06 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease; Hyponatremia; Hypoalbuminemia
MeSH Terms: conditions — Coronary Artery Disease; Hyponatremia; Hypoalbuminemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary artery disease is a common medical disease in many populations. The pathogenesis of this disease is very complex. Surgery is one of the treatment choices. Assessing the risk factors will improve the surgical outcome. In this study some biochemical parameters were evaluated to find out the relationship between these parameters (electrolytes and albumin vs)

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent coronary artery bypass graft surgery
* Elective surgery

Exclusion Criteria:

* Pediatric patients
* Off-pump surgery
* Emergent surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 1157 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
myocardial infarction | One month
  Increase in cardiac enzymes( >0,1 µg/L )

IPD SHARING:
Plan to Share IPD: Undecided